CLINICAL TRIAL: NCT05575154
Title: Is the ISNT Rule Still a Rule : a Study to Determine Prevalence of the ISNT Rule and Its Variants in the Normal Population
Brief Title: ISNT Rule in Normal Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Sayed, Resident ophthalmologist, Assiut University
Other Study IDs: ISNT rule
Record Dates: First submitted 2021-10-09; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma
Keywords: ISNT rule in normal population
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: optical coherence tomography (OCT) — measuring retinal nerve fiber layer and neuroretinal rim thickness

SUMMARY:
This study sought to determine the percentage of normal eyes that followed the ISNT rule by retinal nerve fiber layer (RNFL) and neuroretinal rim thickness measurements using optical coherence tomography (OCT) , and secondarily, whether alternative rules may be more applicable or easily generalized.

DETAILED DESCRIPTION:
Glaucoma is a disease of the optic nerve, which results in structural optic nerve head (ONH) damage and functional visual field (VF) loss. It has increased as a cause of global blindness from 4.4% in 1990 to 6.3% in 2010. Its global prevalence is also increasing from 3.54% or 64.3 million people in 2013 to a projected 111.8 million people by 2040. Detection of structural ONH damage is critical for early diagnosis, because ONH changes usually precede VF loss. Two cornerstone elements of the ONH and peripapillary examination are stereo disc photography and optical coherence tomography (OCT) retinal nerve fiber layer (RNFL) thickness measurements. By analyzing the neuroretinal rim in disc photos of normal subjects, Jonas et al found that the rim width typically exhibited a specific pattern of the inferior (I) rim being the widest, followed by the superior (S) rim, then the nasal (N) rim, and then the temporal (T) rim being the thinnest. This specific neuroretinal rim pattern was later coined by Elliot Werner as the "ISNT rule." Because neuroretinal rim loss is a hallmark feature of glaucoma, patients who deviate from the ISNT rule may need to be watched more closely for glaucoma. The RNFL, on the other hand, has also been shown in histological studies in normal, non-glaucomatous eyes to exhibit a similar pattern of the inferior quadrant being the thickest, followed by the superior, nasal, then temporal quadrant. Since RNFL thinning, particularly in the superior and inferior quadrants, is also a characteristic structural change in glaucoma, deviation from the ISNT rule for RNFL thickness may also be an early indicator of glaucomatous structural change. Therefore, many investigators have sought to determine whether the ISNT rule, either applied to the neuroretinal rim disc photos or to RNFL thickness measurements, is useful in the diagnosis of glaucoma or not. However, the optic disc photo ISNT rule studies are conflicting, with some finding the ISNT rule and its variants clinically useful, while others have not. In contrast, RNFL ISNT rule studies based on OCT findings are in uniform agreement, stating that the ISNT rule and its variants were not helpful in the diagnosis of glaucoma. Some have hypothesized that the ISNT rule is not easily generalizable to the individual, because the initial studies were derived from mean values. Therefore, some of the limitations of the ISNT rule may stem from the fact that it is unclear what percentage of individual normal eyes follow the ISNT rule. Other limitations may arise from the fact that perhaps other rules may be more common in the normal population.

ELIGIBILITY:
Inclusion Criteria:

* a normal eye examination without ocular diseases except for cataracts
* best corrected vision of > 6/12
* a normal VF test result defined by a pattern standard deviation value of > 5% compared to age matched controls in the perimeter's normative database and a glaucoma hemifield test within normal limits
* a spherical equivalent of between -5 and +5 diopters.

Exclusion Criteria:

* unreliable VF testing with > 33% fixation losses, > 20% false positives, or > 20% false negatives.
* any history of ocular hypertension or intraocular pressures > 21mmHg at the time of the visit;
* inter-eye cup-to-disc ratio (CDR) asymmetry of > 0.2;CDR of > 0.4
* history of a neurologic disease or systemic medication that could produce VF defects.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Normal population
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
ISNT rule prevalence in normal population | Baseline
  the percentage of normal eyes that followed the ISNT rule by retinal nerve fiber layer and neuroretinal rim thickness measurements using (OCT)

SECONDARY OUTCOMES:
variants of ISNT rule | Baseline
  whether alternative rules may be more applicable or easily generalized than the ISNT rule like IS,IST, TSINT rule .

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elnasser A Mohamed, PhD, Study Director — Assiut University

REFERENCES:
- [Background] Foster PJ, Buhrmann R, Quigley HA, Johnson GJ. The definition and classification of glaucoma in prevalence surveys. Br J Ophthalmol. 2002 Feb;86(2):238-42. doi: 10.1136/bjo.86.2.238. PMID 11815354
- [Background] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Background] Bourne RR, Taylor HR, Flaxman SR, Keeffe J, Leasher J, Naidoo K, Pesudovs K, White RA, Wong TY, Resnikoff S, Jonas JB; Vision Loss Expert Group of the Global Burden of Disease Study. Number of People Blind or Visually Impaired by Glaucoma Worldwide and in World Regions 1990 - 2010: A Meta-Analysis. PLoS One. 2016 Oct 20;11(10):e0162229. doi: 10.1371/journal.pone.0162229. eCollection 2016. PMID 27764086
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Keltner JL, Johnson CA, Anderson DR, Levine RA, Fan J, Cello KE, Quigley HA, Budenz DL, Parrish RK, Kass MA, Gordon MO; Ocular Hypertension Treatment Study Group. The association between glaucomatous visual fields and optic nerve head features in the Ocular Hypertension Treatment Study. Ophthalmology. 2006 Sep;113(9):1603-12. doi: 10.1016/j.ophtha.2006.05.061. PMID 16949445
- [Background] Broadway DC, Nicolela MT, Drance SM. Optic disk appearances in primary open-angle glaucoma. Surv Ophthalmol. 1999 Jun;43 Suppl 1:S223-43. doi: 10.1016/s0039-6257(99)00007-7. PMID 10416767
- [Background] Jonas JB, Budde WM. Diagnosis and pathogenesis of glaucomatous optic neuropathy: morphological aspects. Prog Retin Eye Res. 2000 Jan;19(1):1-40. doi: 10.1016/s1350-9462(99)00002-6. PMID 10614679
- [Background] Jonas JB, Gusek GC, Naumann GO. Optic disc, cup and neuroretinal rim size, configuration and correlations in normal eyes. Invest Ophthalmol Vis Sci. 1988 Jul;29(7):1151-8. PMID 3417404
- [Background] Jonas JB, Budde WM, Panda-Jonas S. Ophthalmoscopic evaluation of the optic nerve head. Surv Ophthalmol. 1999 Jan-Feb;43(4):293-320. doi: 10.1016/s0039-6257(98)00049-6. PMID 10025513
- [Background] Varma R, Skaf M, Barron E. Retinal nerve fiber layer thickness in normal human eyes. Ophthalmology. 1996 Dec;103(12):2114-9. doi: 10.1016/s0161-6420(96)30381-3. PMID 9003346
- [Background] Dichtl A, Jonas JB, Naumann GO. Retinal nerve fiber layer thickness in human eyes. Graefes Arch Clin Exp Ophthalmol. 1999 Jun;237(6):474-9. doi: 10.1007/s004170050264. PMID 10379607
- [Background] Jonas JB, Budde WM, Lang P. Neuroretinal rim width ratios in morphological glaucoma diagnosis. Br J Ophthalmol. 1998 Dec;82(12):1366-71. doi: 10.1136/bjo.82.12.1366. PMID 9930265
- [Background] Harizman N, Oliveira C, Chiang A, Tello C, Marmor M, Ritch R, Liebmann JM. The ISNT rule and differentiation of normal from glaucomatous eyes. Arch Ophthalmol. 2006 Nov;124(11):1579-83. doi: 10.1001/archopht.124.11.1579. PMID 17102005
- [Background] Law SK, Kornmann HL, Nilforushan N, Moghimi S, Caprioli J. Evaluation of the "IS" Rule to Differentiate Glaucomatous Eyes From Normal. J Glaucoma. 2016 Jan;25(1):27-32. doi: 10.1097/IJG.0000000000000072. PMID 24844540
- [Background] Morgan JE, Bourtsoukli I, Rajkumar KN, Ansari E, Cunliffe IA, North RV, Wild JM. The accuracy of the inferior>superior>nasal>temporal neuroretinal rim area rule for diagnosing glaucomatous optic disc damage. Ophthalmology. 2012 Apr;119(4):723-30. doi: 10.1016/j.ophtha.2011.10.004. Epub 2012 Feb 24. PMID 22365059
- [Background] Dave P, Shah J. Applicability of ISNT and IST rules to the retinal nerve fibre layer using spectral domain optical coherence tomography in early glaucoma. Br J Ophthalmol. 2015 Dec;99(12):1713-7. doi: 10.1136/bjophthalmol-2014-306331. Epub 2015 May 28. PMID 26021327
- [Background] Pradhan ZS, Braganza A, Abraham LM. Does the ISNT Rule Apply to the Retinal Nerve Fiber Layer? J Glaucoma. 2016 Jan;25(1):e1-4. doi: 10.1097/IJG.0000000000000064. PMID 24777047
- [Background] Sihota R, Srinivasan G, Dada T, Gupta V, Ghate D, Sharma A. Is the ISNT rule violated in early primary open-angle glaucoma--a scanning laser tomography study. Eye (Lond). 2008 Jun;22(6):819-24. doi: 10.1038/sj.eye.6702798. Epub 2007 Apr 13. PMID 17435693